CLINICAL TRIAL: NCT06760260
Title: A Study to Evaluate the Safety and Efficacy of CI-135 CAR-T Cell Injection in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Evaluation of the Safety and Efficacy of Human CI-135 (FLT3) Targeted CAR-T Cells Injection for Subjects with Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-AML02-POC
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Anti CI-135 (FLT3) CAR-T Injection (Experimental): Single administration: 0.5 * 10^6 CAR-T cells/kg, 1.0 * 10^6 CAR-T cells/kg
  Interventions: Drug: Human Derived anti-CI135 CAR-T Injection

INTERVENTIONS:
Drug: Human Derived anti-CI135 CAR-T Injection — Autologous genetically modified anti-CI135 CAR transduced T cells
  Other Names: FLT3 CAR-T

SUMMARY:
This study is a single-arm, open-label, dose-escalating trial to explore the safety, tolerability and pharmacokinetic/pharmacodynamics characteristics of anti human CI-135 (FLT3) CAR-T Injection , and to preliminarily observe the efficacy of the trial drug in patients with relapsed/refractory Acute Myeloid Leukemia.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

* Subjects volunteer to participate in clinical trails, understand and inform the trials and sign informed consent form, be willing to complete all the trial procedures;
* Aged from 18 to 70 years (including cut-off value), Male and female;
* Expected survival > 12 weeks;
* Previously diagnosed as Acute Myeloid Leukemia by ELN updated criteria (2017) and one of the following indicators that is satisfied:

  1. AML patients who have not achieved complete remission (CR) after at least three cycles of standard induction therapy, or
  2. AML patients who achieved complete remission after induction therapy but relapsed within one year, or
  3. AML patients who achieved complete remission after induction therapy for more than one year but did not achieve remission after one cycle of chemotherapy with the original regimen following relapse, or
  4. AML patients who relapsed after transplantation, or
  5. AML patients who experienced two or more relapses. Note: For patients meeting conditions a), b), or c) with FLT3 mutations, they must have undergone at least one treatment with a tyrosine kinase inhibitor (TKI) without achieving complete remission or have relapsed after achieving complete remission, except for those who cannot tolerate TKI therapy or have contraindications to TKI treatment.
* Positive for FLT3 mutation confirmed by leukemia cell genetic testing, or FLT3 expression ≥35%;
* ECOG performance status score of 1-2;
* Liver, kidney, heart, and lung functions meeting the following criteria:

  1. Glomerular filtration rate (GFR) ≥60 ml/min/1.73 m² or serum creatinine ≤2 times the upper limit of normal (ULN);
  2. Serum AST and ALT ≤3 times of ULN, and total bilirubin ≤1.5 times the ULN;
  3. Oxygen saturation > 92%;
  4. Left ventricular ejection fraction (LVEF) ≥50%, with no pericardial effusion observed on ultrasound, and no clinically significant electrocardiographic abnormalities.
* Able to understand the study and sign the informed consent form.

Exclusion Criteria:

* Diagnosed as acute promyelocytic leukemia (APL M3);
* With any presence of other uncontrolled malignancies (unless evaluated as unlikely to interfere with the safety or efficacy assessment of the trial);
* Previously treated with CAR-T cells or other genetically modified cellular therapies
* Displayed history or evidence of significant cardiovascular risks, including any of the following: congestive heart failure, unstable angina, clinically significant arrhythmias (e.g., ventricular fibrillation, ventricular tachycardia), coronary angioplasty within 6 months before administration, implantable cardiac defibrillator, or any clinically relevant comorbidities that pose safety risks or interfere with study assessments, procedures, or completion;
* Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with HBV DNA levels ≥ the detection limit in peripheral blood; positive for hepatitis C virus (HCV) antibody with detectable HCV RNA; positive for human immunodeficiency virus (HIV) antibodies; or positive for syphilis testing;
* Positive for acute or chronic hepatitis C. Exceptions: acute hepatitis C with complete viral clearance; chronic hepatitis C with a sustained virological response (SVR24) 24 weeks post-treatment confirming undetectable viral load;
* Having history of arterial or venous thrombosis within 3 months prior to enrollment;
* Having history of Graft-versus-host disease requiring systemic immunomodulators;
* Having history of central nervous system diseases or conditions requiring treatment (e.g., uncontrolled seizures);
* Having uncontrolled active infections;
* Known allergy to any components of CI-135 CAR-T cell formulation or the lymphodepletion regimen (cyclophosphamide and fludarabine);
* Currently pregnant or lactating female, or female subjects planning pregnancy within 1 year after cell infusion, or male subjects with partners planning pregnancy within 1 year after infusion;
* Having other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | 28 days post infusion
  Safety Indicator

SECONDARY OUTCOMES:
Pharmacokinetics parameters - Maximum CAR level in peripheral blood (Cmax) | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters -Time to maximum CAR level in peripheral blood (Tmax) | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - 28-day Area under Curve of CAR level in peripheral blood (AUC0-28) | 2 years post infusion
  Effectiveness Metrics
Pharmacodynamics characteristics - Cytokines Concentrations, cytokines level in peripheral blood | 2 years post infusion
  Effectiveness Metrics, determined via ELISA, including but not limited to:
  Interleukin-15 (IL-15) by pg/μl blood sample; Interleukin-6 (IL-6) by pg/μl blood sample; Granzyme B by pg/μl blood sample; Interferon-γ (IFN-γ) by pg/μl blood sample; Tumor Necrocis Factor α (TNF-α) by pg/μl blood sample;
Overall Response Rate (ORR) | 28 days post infusion
  ORR defined as proportion of subjects who achieved Partial Remission (PR), Morphologic leukemia-free state (MLFS) or better (CR, CRi) according to the ELN 2017 as determined by an Investigator assessment at day 28.
Progression-free Survival (PFS) | 2 years post infusion
  PFS defined as time from date of initial infusion of CAR-T to date of first disease progression according to ELN2017 criteria, or death due to any cause, whichever occurs first.
Overall Survival (OS) | 2 years post infusion
  OS is measured from the date of the initial infusion of CAR-T to the date of the subject's death.
Duration of Response (DOR) | 2 years post infusion
  DOR will be calculated among responders (PR, MLFS or better) from the date of initial response (PR, MLFS or better) to the date of first documented evidence of progressive disease, as defined in the ELN criteria (2017).

OTHER OUTCOMES:
HAMA Immunogenicity | 2 years post infusion
  Determination of the immunogenicity via human anti-mouse antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China